CLINICAL TRIAL: NCT05362396
Title: Inspiratory Muscle Training in Respiratory Capacity, Life Quality, Lumbar Pain, Phase Angle and Body Composition in Patients With Fibromyalgia.
Brief Title: Inspiratory Muscle Training With Powerbreath Device in Patients With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Fibro-UFV22
Record Dates: First submitted 2022-04-21; First posted 2022-05-05 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory muscle training (Experimental): Inspiratory muscle training with Powerbreath IMT device, for a duration of 8 weeks. Treatment as usual
  Interventions: Other: Inspiratory Muscle Training with Powerbreath IMT device.
- No training program (No Intervention): Without inspiratory muscle training. Treatment asusual.

INTERVENTIONS:
Other: Inspiratory Muscle Training with Powerbreath IMT device. — Inspiratory muscle training with Powerbreath IMT device, for a duration of 8 weeks. Each day, each subject perform 5 sets of 10 repetitions, 5 days a week. The endurance of the device increases along the study, initiating with the 50% of their own maximum inspiratory pressure (MIP) during the first week, 2nd week: 55% MIP, 3rd week: 60% MIP, 4th week: 65% MIP, 5th week: 70% MIP, 6th week: 75% MIP, 7th week: 80% MIP and 8th week:80% MIP
  Arms: Inspiratory muscle training

SUMMARY:
Context/background: people affected by fibromyalgia see their own life totally disturbed after the diagnosis. This disease also courses, apart from the functional and depressing worsening, with internal damage manifested by a cardio respiratory deterioration. There are not many clinical studies publications about this disease given that is considered a weird illness with short prognosis.

Objectives: to examine the effects of the inspiratory muscle training (IMT) on respiratory muscle strength, lumbar pain, quality of life, phase angle and body composition in patients with Fibromyalgia.

The participants of experimental group will conduct 5 sets of 10 inspirations per day, 5 days per week, through 8 weeks.

DETAILED DESCRIPTION:
Methods: 40 volunteer patients, female, with fibromyalgia will take part of the cuasi-experimental study and they will be divided into two groups: an experimental group (n = 20) and a control group (n = 20). The Maximum Inspiratory Pressure (PIM), the quality of life, lumbar pain, phase angle and body composition will be measured.

Inspiratory muscle training with Powerbreath IMT device, for a duration of 8 weeks. Each day, each subject perform 5 sets of 10 inspirations, 5 days a week. The endurance of the device increases along the study, initiating with the 50% of their own maximum inspiratory pressure (MIP) during the first week, 2nd week: 55% MIP, 3rd week: 60% MIP, 4th week: 65% MIP, 5th week: 70% MIP, 6th week: 75% MIP, 7th week: 80% MIP and 8th week:80% MIP

After 8 weeks, all participants will fill up again all scales and post training measurements will be taken.

ELIGIBILITY:
Inclusion Criteria:

* subjects with fibromyalgia

Exclusion Criteria:

-

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
MIP | Change from baseline inspiratory muscle strength at 8 weeks]
  Maximum Inspiratory Pressure. Inspiratory muscle strength will be measured in % by a POWER-breathe device
Pain: Pressure algometry | 8 week
  Pain will be measured with pressure algometry measured in Kg from 0 to 5kg.
Pain :VAS | change from baseline after 8 week
  Visual Analogic Scale. Pain will be measured with a visual analog scale from 0 to 10. 0 points is no pain.
phase angle | 8 week
  The phase angle, which is measured via bioelectrical impedance analysis (BIA), InBody 770 ,is a clinically important bioimpedance parameter used for nutritional assessment and evaluating the risk of various diseases. The phase angle was calculated automatically by the BIA device from these two components according to the following formula: phase angle (°) = (reactance/resistance) × (180°/π).
Fibromyalgia Impact Questionnaire (S-FIQ) | 8 week
  The Fibromyalgia Impact Questionnaire (FIQ) is a brief 10-item, self-administered instrument that measures physical functioning, work status, depression, anxiety, sleep, pain, stiffness, fatigue, and well being. The total FIQ score is between 0-100. Thus, 0 represents the highest functional capacity and quality of life and 100 the worst state.
Diaphragm tickness | Change from baseline diaphragm muscle thickness at 8 weeks
  Diaphragm muscle thickness will be measured in mm by an ultrasound device

CONTACTS AND LOCATIONS:
Overall Officials: Davinia Vicente Campos, PhD, Principal Investigator — Universidad Francisco de Vitoria
Locations (1):
- Universidad Francisco de Vitoria, Pozuelo de Alarcón, Madrid, Spain